CLINICAL TRIAL: NCT07006519
Title: The Prevalence of Incisal Angle of Maxillary Central Incisors in Adults: A Cross-sectional Study
Brief Title: The Prevalence of Incisal Angle of Maxillary Central Incisors in Adults
Status: Not yet recruiting | Type: Observational
Sponsor: Misr International University (Other)
Responsible Party: Principal Investigator, Ahmed Abo El Futtouh, Exectutive and Clinical director of Implantology Master program, MIU, Misr International University
Other Study IDs: IDCE 15
Record Dates: First submitted 2025-05-04; First posted 2025-06-05 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Anterior Teeth
Keywords: anterior teeth; central incisor

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Central Incisors: intra-oral scan for central incisors

SUMMARY:
This study is to assess the prevalence of different incisal angle of maxillary central incisors in a sample of adults.Materials and methods: The current study will include 300 sound natural maxillary central incisor. intraoral scan will be taken for all cases to measure the incisal angle.

DETAILED DESCRIPTION:
This study is aimed to assess the prevalence of different incisal angle of maxillary central incisors in a sample of adults population with sound anterior central incisors. The current study will include 300 sound natural maxillary central incisor. For each, an intraoral scan will be taken to measure the incisal angle. , wither having a mesial or distal incisal angle and its degree and how frequent each one. the scans will be aligned in same xyz axis for proper standardization for the measurements.

ELIGIBILITY:
Inclusion Criteria:

* sound natural teeth

Exclusion Criteria:

* rotated teeth
* pathological migration of teeth
* patients subjected to trauma for anterior teeth

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult individuals with sound central incisor
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2026-03-15 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Incisal angle | Baseline
  Incisal angle of central incisors will be measured on Medit computer software from scanned STL files. Each angle will be measured in degrees

CONTACTS AND LOCATIONS:
Locations (1):
- International Dental Clinic Educational centre, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided